CLINICAL TRIAL: NCT01153191
Title: Developing Evidence of Effectiveness for Adjuvant Interventions Designed to Minimize Surgical Site Infections
Brief Title: Effectiveness for Interventions to Minimize Surgical Site Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas Anthony, MD, Dallas VA Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: #10-046
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Infections
Keywords: colorectal surgery
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressurized irrigation (Experimental): first group-After closure of patients abdominal wall fascia, Hydrostatic irrigation with 3 liters of normal saline with Simpulse Solo irrigation system (Davol) at less than 15PSI will be applied to subcutaneous tissues prior to closure
  Interventions: Procedure: Normal saline pressurized irrigation
- Sub Q Antibiotic (Experimental): second group of patients will receive 2mg/lg of gentamicin in 20 ml of sterile saline injected into the superficial tissues above the ABD wall fascia prior to initial incision
  Interventions: Drug: sub-q gentamicin

INTERVENTIONS:
Procedure: Normal saline pressurized irrigation — same
  Other Names: 1st group
  Arms: Pressurized irrigation
Drug: sub-q gentamicin — 2mg/kg of gentamicin in 20 ml of sterile saline up to max dose of 120mg injected above the abdominal wall fascia- the length of the incision will be marked and injection made with intent being to evenly distribute the volume of injection in the subcutaneous tissues in immediate vicinity of and prior to the initial incision- analogous to the technique employed when using local anesthetic
  Other Names: 2nd group
  Arms: Sub Q Antibiotic

SUMMARY:
The purpose of this study is to evaluate two different simple and inexpensive extra treatments during colorectal surgeries to see if this will reduce the rate of post operative infections

DETAILED DESCRIPTION:
The population for inclusion for this study will be drawn from the patients undergoing elective transabdominal colorectal surgery. This population was chosen due to its inherently high rate of superficial-incisional infection.Colorectal procedures stand out as a particularly highrisk surgery with respect to SSI. Several studies have reported rates of infection of 25% or more making colorectal surgeries an excellent opportunity for testing new strategies to reduce SSI.

This pilot project seeks to preliminarily evaluate two new strategies that are inexpensive and could be readily incorporated into current practice. The strategies are pressurized irrigation of the superficial surgical wound (above the fascia) and subcutaneous injection of gentamicin into the surgical wound prior to initial skin incision. Comparison will be made between prospectively enrolled patients and historic controls.The hypothesis to be tested is that these interventions will significantly reduce superficial incisional infection rates compared with historic control.

ELIGIBILITY:
Inclusion Criteria:

* VA patients getting transabdominal,elective colorectal procedures
* willing and capable of giving self informed consent

Exclusion Criteria:

* patients unable to give informed consent
* emergency colorectal procedures
* transanal procedures
* patients who have contaminated or dirty wounds that would preclude attempts at skin closure at the conclusion of the procedure
* patients undergoing appendectomy
* patients undergoing intraabdominal procedures not including surgical resection of the colon or rectum (ie.procedures involving small bowel , stomach)
* patients with pre/op creatinine clearance less than 20ml/min
* patients with known allergy or hypersensitivity to gentamicin
* patients that have received gentamicin within 2 weeks of potential study date

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Infection rate in colorectal surgeries in each of two treatment arms as compared to historic controls | 30 days after surgery
  pilot study to evaluate 1. pressurized irrigation of the superficial surgical wound after fascial closure in 40 patients and 2. subcutaneous gentamicin into the surgical area prior to initial incision in 40 patients and compare rates of surgical site infections after 30 days to historic controls.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Dineen, MD, Principal Investigator — VANTXHCS
Locations (1):
- VANTXHCS, Dallas, Texas, United States

REFERENCES:
- [Derived] Dineen SP, Pham TH, Murray BW, Parker BJ, Hartless K, Anthony T, Huerta S. Feasibility of subcutaneous gentamicin and pressurized irrigation as adjuvant strategies to reduce surgical site infection in colorectal surgery: results of a pilot study. Am Surg. 2015 Jun;81(6):573-9. PMID 26031269